CLINICAL TRIAL: NCT02384551
Title: Dietary Carbohydrate Effects on GERD in Obese Veterans: Nutritional or Hormonal?
Brief Title: Dietary Carbohydrate and GERD in Veterans
Acronym: DietGERD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLNB-006-14S
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Gastroesophageal Reflux Disease; Obesity
Keywords: GERD; diet; carbohydrate; obesity
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity | interventions — Dietary Carbohydrates

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- HTHS (Active Comparator): High total carbohydrate with high total simple carbohydrate diet
  Interventions: Other: Dietary Carbohydrate
- HTLS (Experimental): High total carbohydrate with low total simple carbohydrate diet
  Interventions: Other: Dietary Carbohydrate
- LTHS (Experimental): Low total carbohydrate with high total simple carbohydrate diet
  Interventions: Other: Dietary Carbohydrate
- LTLS (Experimental): Low total carbohydrate with low total simple carbohydrate diet
  Interventions: Other: Dietary Carbohydrate

INTERVENTIONS:
Other: Dietary Carbohydrate — 9 week menu of dietary carbohydrate modification

SUMMARY:
4-Arm Diet Intervention Investigating Effects of Dietary Carbohydrate Type and Amount on gastroesophageal pH, gastroesophageal reflux disease (GERD) symptoms and medication use.

DETAILED DESCRIPTION:
delayed due to COVID related research shutdown

Specific Hypothesis: The preliminary findings suggest a physiological mechanism between dietary intake and GERD that may be related to type of dietary carbohydrate intake (complex vs simple carbohydrate). The investigators hypothesize that modifying the type of dietary carbohydrate consumed - by reducing the proportion of simple carbohydrate (sugars) consumed - will reduce or resolve GERD symptoms and medication use in obese Veterans with chronic GERD. The investigators further hypothesize that the mechanistic effects of reducing simple carbohydrate intake is related to either: a) improved dietary fiber intake and/or glycemic load, and thus, reduced amount and duration of esophageal acid exposure; and/or b) improved insulin sensitivity which would positively influence the function of key gastrointestinal hormones (ie, gastrin, glucagon, GLP-1, ghrelin11) that regulate gastric motility and/or lower esophageal sphincter function.

Aim 1: To determine effects of dietary carbohydrate consumed (amount and type) on percent time with esophageal pH < 4.0, as well as number of reflux episodes, GERD symptoms and GERD medication use, in 200 obese Veterans who have chronic high frequency of GERD symptoms. To meet this aim the investigators will use a randomized controlled trial in which the investigators manipulate amount of total and simple dietary carbohydrate intake for duration of 9 weeks.

Aim 2: To assess associations between GERD resolution variables and factors related to potential mechanisms by which modifying dietary carbohydrate intake could resolve/reduce GERD in obese Veterans.

2a: The investigators will investigate associations related to whether the effect is nutritionally mediated by measuring change in dietary fiber load and dietary glycemic load, and thus, whether these changes are related to improved gastric acid secretion (% time pH < 4), gastric motility, and/or the other parameters that comprise the Johnson-DeMeester score.

2b: The investigators will also investigate whether effects are associated with changes in the hormonal milieu by measuring hormonal response of gastrin, glucagon, glucagon-like peptide-1 (GLP-1), ghrelin and insulin, which could potentially influence gastric acid secretion, gastric motility and/or lower esophageal sphincter function.

ELIGIBILITY:
Inclusion Criteria:

Age 21 or over BMI 30-39.9 GERD

Exclusion Criteria:

* History of type 1 diabetes
* Hernia or strictures
* Gastroparesis
* Extra-esophageal GERD
* Barrett's esophagus or Esophageal adenocarcinoma
* History of gastric or bariatric or esophageal surgery, radiation or cancer
* History of gastrointestinal malabsorption
* Alcohol averaging > 2 drinks per day during past 3 months
* Pregnancy / Lactation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Niswender, MD PhD, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (1):
- Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Data will be provided as group data upon publication

REFERENCES:
- [Result] Gu C, Olszewski T, King KL, Vaezi MF, Niswender KD, Silver HJ. The Effects of Modifying Amount and Type of Dietary Carbohydrate on Esophageal Acid Exposure Time and Esophageal Reflux Symptoms: A Randomized Controlled Trial. Am J Gastroenterol. 2022 Oct 1;117(10):1655-1667. doi: 10.14309/ajg.0000000000001889. Epub 2022 Jun 21. PMID 35973185

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HTHS | HTLS | LTHS | LTLS
Started | 35 | 40 | 36 | 39
Completed | 22 | 26 | 22 | 25
Not Completed | 13 | 14 | 14 | 14
Not completed — Lost to Follow-up | 13 | 14 | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HTHS | HTLS | LTHS | LTLS | Total
Number analyzed (Participants) | 22 | 26 | 22 | 25 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 26 | 22 | 25 | 95
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (11.1) | 58.4 (15.3) | 56.0 (12.8) | 59.9 (10.6) | 59.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 6 | 15
  Male | 19 | 23 | 19 | 19 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 14 | 11 | 14 | 50
  White | 11 | 12 | 11 | 11 | 45
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 26 | 22 | 25 | 95

OUTCOME MEASURES:

1. Primary Outcome: Gastroesophageal pH
Description: ambulatory ph monitoring for percent time gastroesophageal ph < 4 in 24 hrs
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: percent time ph < 4 in 24 hrs
Arm/Group | HTHS | HTLS | LTHS | LTLS
Number analyzed (Participants) | 22 | 26 | 22 | 25
percent time ph < 4 in 24 hrs | 7.3 (12.1) | 6.6 (8.4) | 3.7 (4.2) | 4.9 (4.7)

2. Secondary Outcome: Gastroesophageal Reflux Disease Questionnaire (GERDQ) Score
Description: GERD symptoms using Gastroesophageal Reflux Disease Questionnaire (GERDQ) Score, score is based on a scale, from 0-18, with higher score indicating more symptoms. There is not a measure of central tendency, just the total score as reported.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: final score
Arm/Group | HTHS | HTLS | LTHS | LTLS
Number analyzed (Participants) | 22 | 26 | 22 | 25
final score | 5.1 (3.8) | 3.2 (3.1) | 4.5 (4.5) | 3.5 (2.9)

3. Secondary Outcome: Gastroesophageal Scale Assessment Symptom (GSAS) Score
Description: GERD symptoms measured as Gastroesophageal Scale Assessment Symptom (GSAS) score. Scores range from 0-45, with higher scores indicating more symptoms. Not a measure of central tendency.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: total score
Arm/Group | HTHS | HTLS | LTHS | LTLS
Number analyzed (Participants) | 22 | 26 | 22 | 25
total score | 5.6 (2.4) | 4.1 (2.0) | 5.6 (2.3) | 4.5 (2.1)

ADVERSE EVENTS:
Time Frame: 9 weeks
Description: no difference
Arm/Group | HTHS | HTLS | LTHS | LTLS
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/40 | 0/36 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/40 | 0/36 | 0/39
Other Adverse Events (participants affected / at risk) | 0/35 | 0/40 | 0/36 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HTHS (N=35) | HTLS (N=40) | LTHS (N=36) | LTLS (N=39)
pill stuck in throat (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT02384551/Prot_SAP_000.pdf
  • Informed Consent Form (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT02384551/ICF_001.pdf